CLINICAL TRIAL: NCT01805180
Title: A Controlled Evaluation of the Spectra Optia® Apheresis System's Granulocyte / Polymorphonuclear (PMN) Cell Collection Procedure
Brief Title: Evaluation of the Spectra Optia PMN Cell Collection Procedure
Acronym: PMNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CTS-5010
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-02

CONDITIONS: Granulocyte/ Polymorphonuclear Cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Spectra Optia followed by COBE Spectra (Other): Controlled evaluation of Granulocyte/Polymorphonuclear Cell Collection on the Spectra Optia device followed by the COBE Spectra device.
  Interventions: Device: Granulocyte/Polymorphonuclear Cell Collection (COBE Spectra System); Device: Granulocyte/Polymorphonuclear Cell Collection (Spectra Optia System)
- Arm 2: COBE Spectra followed by Spectra Optia (Other): Controlled evaluation of Granulocyte/Polymorphonuclear Cell Collection on the COBE Spectra device followed by Spectra Optia.
  Interventions: Device: Granulocyte/Polymorphonuclear Cell Collection (COBE Spectra System); Device: Granulocyte/Polymorphonuclear Cell Collection (Spectra Optia System)

INTERVENTIONS:
Device: Granulocyte/Polymorphonuclear Cell Collection (COBE Spectra System) — In Arm 1 the first PMN cell collection will be performed using the Spectra Optia System and the second PMN cell collection using the COBE Spectra System.
Device: Granulocyte/Polymorphonuclear Cell Collection (Spectra Optia System) — In Arm 2 the first PMN cell collection will be performed using the COBE Spectra System and the second PMN cell collection using the Spectra Optia System.

SUMMARY:
The purpose of this study is to compare the procedures for the collection PMN cells on Terumo BCT's Spectra Optia® and COBE® Spectra Apheresis Systems.

DETAILED DESCRIPTION:
The purpose of this study is to compare the procedures for the collection of granulocyte/ polymorphonuclear (PMN) cells on Terumo BCT's Spectra Optia® and COBE® Spectra Apheresis Systems and to establish the non-inferiority of the Spectra Optia Apheresis System with respect to the primary study endpoint, granulocyte/PMN cell collection efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable health status and vital signs per the AABB blood donation guidelines to permit blood donation, including:

  1. Blood pressure ≥ 90/50 and ≤ 200/120 mmHg,
  2. Pulse > 40 and < 100 beats/min, and
  3. Temperature < 99.5ºFahrenheit (F).
* Able to read, understand, and sign an English informed consent form.
* Age ≥ 18 years.
* Weight ≥ 50kg and < 227kg.
* Male or non-pregnant, non-nursing female (a negative serum pregnancy test at screening and a negative urine pregnancy test prior to each mobilization).
* Acceptable screening laboratory test results prior to the first PMN cell mobilization, including:

  1. WBC count in the range: 3,500-10,800/uL,
  2. Hematocrit in the range: 38-65%,
  3. Platelet count in the range: 150,000-400,000/uL,
  4. Coagulation tests: PT not greater than 1.1 times the upper limit of the local laboratory reference range; PTT not greater than 1.2 times the upper limit of the local laboratory reference range,
  5. Serum electrolyte concentrations: potassium in the range 3.6-5.1 mmol/L; calcium in the range 8.5-10.3 mg/dL,
  6. Serum creatinine not greater than 1.5mg/dL, and
  7. ALT not greater than 1.5 times the upper limit of the local laboratory reference range. *** Up to two (2) of the above screening laboratory test results may fall outside of these ranges, if in the judgment of the principal investigator or designee, they do not constitute a significant risk to the subject. Any excused deviations from the above will be listed and summarized with the final report.***
* Adequate dual peripheral venous access to allow collection of granulocytes (PMN cells) and return of remaining cells, platelets and plasma.
* If male, willing to use a condom during sexual relations with a female partner of child bearing potential until 48 hours following each G-CSF injection.
* If female, willing to use a medically-acceptable contraceptive until 48 hours following each G-CSF injection.

Exclusion Criteria:

* Positive screening for any of the following: HIV, HBV (except isolated HB core Ab reactivity), HCV, HTLV, Syphilis or West Nile Virus.
* Currently pregnant or breast-feeding.
* Collection or loss of specific volumes of whole blood or blood components during specified timeframes:

  1. more than 550mL of whole blood within the prior 56 days, or
  2. more than 3L of whole blood or 1.5L of red blood cells within the prior 12 months, or
  3. more than 12L of plasma within the prior 12 months, or
  4. a leukapheresis within the prior six weeks, or
  5. a plateletpheresis within the prior 48 hours or two within the prior 7 days or twenty-four within the last 12 months, or
  6. a plasmapheresis within the prior 48 hours or two within the prior 7 days.
* History of congestive heart failure.
* History of uncontrolled hypertension (SBP/DBP >200/120 mmHg).
* History or suspicion of active, peptic ulcer disease.
* History of diabetes mellitus.
* History of hematologic malignancy or chronic hematologic disorder.
* Family history (parents, siblings, children) of hematologic malignancy.
* History of deep vein thrombosis or venous thromboembolism, or bleeding disorder.
* History of sickle cell disease or a positive SickleDex screen.
* History of iritis or episcleritis.
* History of autoimmune condition or disorder, unless approved by principal investigator.
* Presence of psychological traits, or physiological or medical conditions that, in the opinion of the investigator, would make the subject unlikely to tolerate the procedures or complete the study.
* History of use/anticipated need for lithium.
* Received a G-CSF injection in the prior 4 months.
* Known hypersensitivity to ethylene oxide.
* Known hypersensitivity to G-CSF or hypersensitivity to any E. coli-derived products.
* Known hypersensitivity to HES or corn.
* Concurrent participation in another clinical trial or participation in a clinical trial within the past 30 days.
* Subject is being treated with calcium channel blockers and/or antiepileptic medications. Note: This applies only to Subjects at Bonfils Blood Center whose collected product will undergo neutrophil function testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Goodrich, Ph.D, Study Director — Terumo BCT
Locations (3):
- United States (3):
  - Bonfils Blood Center, Denver, Colorado
  - Hoxworth Blood Center, Cincinnati, Ohio
  - Blood Centers of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the specialized donor population of blood centers from February 2013 - July 2013.
Pre-assignment Details: A screening period was used to evaluate and confirm eligibility criteria prior to enrollment & randomization to treatment assignment (Arm 1 or Arm 2). Fifty subjects consented to the pivotal study. Eight pivotal subjects consented but screen failed prior to treatment assignment. Forty-two received treatment assignment below.
Groups:
- Lead-in Donor: Subjects screened and enrolled for the purpose of training on the investigational procedure only. Included in safety analysis only.
- Arm 1 - Spectra Optia Followed by COBE Spectra PMN: Healthy donors who were consented to participate in the pivotal trial and were randomized to receive the PMN collection procedure on the Spectra Optia first, followed by the COBE Spectra.
- Arm 2 - COBE Spectra Followed by Spectra Optia PMN: Healthy donors who were consented to participate in the pivotal trial and were randomized to receive the PMN collection procedure on the COBE Spectra first, followed by the Spectra Optia.
Period: Lead-in Donor Phase
Arm/Group | Lead-in Donor | Arm 1 - Spectra Optia Followed by COBE Spectra PMN | Arm 2 - COBE Spectra Followed by Spectra Optia PMN
Started | 7 | 0 (pivotal trial subjects were not screened or enrolled in this period.) | 0 (pivotal trial subjects were not screened or enrolled in this period.)
Completed | 6 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — screen failure | 1 | 0 | 0
Period: Pivotal Randomization Through Study Exit
Arm/Group | Lead-in Donor | Arm 1 - Spectra Optia Followed by COBE Spectra PMN | Arm 2 - COBE Spectra Followed by Spectra Optia PMN
Started | 0 (lead-in donors were not randomized and did not participate in this period.) | 22 | 20
Completed | 0 | 17 | 15
Not Completed | 0 | 5 | 5

BASELINE CHARACTERISTICS:
Population: Subjects in the Full Set Analysis (n=32) were randomized to either Arm 1 or Arm 2 and completed both procedures as assigned. Subjects who did not complete the collection (withdrawn n=10) did not have data and could not be included in the full set analysis.
Groups:
- Arm 1: In Arm 1 the first PMN cell collection was performed using the Spectra Optia System and the second PMN cell collection using the COBE Spectra System for each subject.
- Arm 2: In Arm 2 the first PMN cell collection was performed using the COBE Spectra System and the second PMN cell collection using the Spectra Optia System for each subject.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (10.99) | 38.3 (13.69) | 36.3 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 8 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 13 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Granulocyte/PMN Cell Collection Efficiency
Description: The primary endpoint is the granulocyte/PMN cell collection efficiency (CE) associated with the Granulocyte (PMN) Collection Procedures on the Spectra Optia and COBE Spectra Apheresis Systems. CE is a measurement of device performance calculated using donor and blood product blood counts collected immediately before and after the PMN collection procedure.
Time Frame: within 1 hour prior and within 5 minutes after each collection procedure
Measure: Mean (Standard Deviation); unit: percent cells processed
Groups:
- Arm 1 - Spectra Optia Followed by COBE Spectra: In Arm 1 the first PMN cell collection was performed using the Spectra Optia System and the second PMN cell collection using the COBE Spectra System for each subject.
- Arm 2 - COBE Spectra Followed by Spectra Optia: In Arm 2 the first PMN cell collection was performed using the COBE Spectra System and the second PMN cell collection using the Spectra Optia System for each subject.
Arm/Group | Arm 1 - Spectra Optia Followed by COBE Spectra | Arm 2 - COBE Spectra Followed by Spectra Optia
Number analyzed (Participants) | 17 | 15
percent cells processed
  Spectra Optia CE% | 54.7 (6.46) | 52.4 (7.43)
  COBE Spectra CE% | 41.9 (6.14) | 44.7 (6.18)

2. Secondary Outcome: Performance
Description: Comparison of collection efficiencies associated with the Granulocyte Cell Collection Procedures on the Spectra Optia and COBE Spectra Apheresis Systems for white blood cells and platelets. CE is a measurement of device performance calculated using donor and blood product blood counts collected immediately before and after the collection procedure.
Time Frame: within 1 hour prior and within 5 minutes after each collection procedure
Measure: Mean (Standard Deviation); unit: percent of cells processed
Arm/Group | Arm 1 - Spectra Optia Followed by COBE Spectra | Arm 2 - COBE Spectra Followed by Spectra Optia
Number analyzed (Participants) | 17 | 15
percent of cells processed
  Spectra Optia WBC CE% | 56.6 (6.15) | 55.4 (6.67)
  COBE Spectra WBC CE% | 44.0 (0.06) | 46.9 (5.96)
  Spectra Optia PLT CE% | 11.2 (1.59) | 10.4 (1.19)
  COBE Spectra PLT CE% | 11.7 (3.09) | 9.7 (2.07)

3. Secondary Outcome: Characterization of Blood Product - PMN Cell Yield
Description: Characterization of the collected blood product, specifically total PMN cell yield. This is a measurement of device performance measured by calculating cell counts in samples from the collected blood product.
Time Frame: within 5 minutes after each collection procedure
Measure: Mean (Standard Deviation); unit: cells *10^10
Arm/Group | Arm 1 - Spectra Optia Followed by COBE Spectra | Arm 2 - COBE Spectra Followed by Spectra Optia
Number analyzed (Participants) | 17 | 15
cells *10^10
  Spectra Optia PMN Cell Yield | 1.4 (0.30) | 1.4 (0.34)
  COBE Spectra PMN Cell Yield | 1.1 (0.28) | 1.2 (0.25)

4. Secondary Outcome: Characterization of Blood Product - PMN Cell Yield Per Liter of Blood Processed
Description: Characterization of the collected blood product, specifically PMN cell yield per liter blood processed. This is a measurement of device performance measured by calculating cell counts in samples from the collected blood product and blood processed measured by the device.
Time Frame: within 5 minutes after each collection procedure
Measure: Mean (Standard Deviation); unit: cells *10^10 per L of blood processed
Arm/Group | Arm 1 - Spectra Optia Followed by COBE Spectra | Arm 2 - COBE Spectra Followed by Spectra Optia
Number analyzed (Participants) | 17 | 15
cells *10^10 per L of blood processed
  Spectra Optia PMN Cell Yield per L of Blood Proces | 1.4 (0.30) | 1.4 (0.34)
  COBE Spectra PMN Cell Yield per L of Blood Proc | 1.1 (0.28) | 1.2 (0.25)

5. Secondary Outcome: Characterization of the Blood Product - PMN Cell Viability
Description: Characterization of the collected blood product, specifically PMN cell viability measured by an assay preformed on the collected blood product.
Time Frame: within 5 minutes after collection procedure
Measure: Mean (Standard Deviation); unit: percent of viable cells
Arm/Group | Arm 1 - Spectra Optia Followed by COBE Spectra | Arm 2 - COBE Spectra Followed by Spectra Optia
Number analyzed (Participants) | 17 | 15
percent of viable cells
  Spectra Optia PMN viability | 99.6 (0.22) | 99.6 (0.28)
  COBE Spectra PMN viability | 99.6 (0.34) | 99.2 (1.81)

6. Secondary Outcome: Characterization of the Blood Product - RBC Contamination
Description: Characterization of the collected blood product, specifically red blood cell (RBC) contamination as measured by hematocrit in the collected PMN product.
Time Frame: within 5 minutes after collection procedure
Measure: Mean (Standard Deviation); unit: RBC percent of product volume
Groups:
- Spectra Optia vs COBE Spectra: All 32 subjects received both the Spectra Optia and the COBE Spectra. RBC contamination results via hematocrit in collected product not reported by randomization treatment arms.
Arm/Group | Spectra Optia vs COBE Spectra
Number analyzed (Participants) | 32
RBC percent of product volume
  Spectra Optia Product HCT | 7.4 (2.62)
  COBE Spectra Product HCT | 7.5 (3.71)

7. Secondary Outcome: Characterization of the Blood Product - Volume
Description: Characterization of the collected blood product, specifically product volume.
Time Frame: within 5 minutes after collection procedure
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Arm 1 - Spectra Optia Followed by COBE Spectra | Arm 2 - COBE Spectra Followed by Spectra Optia
Number analyzed (Participants) | 17 | 15
mL
  Spectra Optia Product Volume | 472.6 (1.77) | 471.9 (1.49)
  COBE Spectra Product Volume | 329.7 (55.72) | 298.5 (53.04)

8. Secondary Outcome: Usability/Assessment of System Operation - Time
Description: Procedure time for collections on the Spectra Optia vs. the COBE Spectra.
Time Frame: Result captured immediately upon completion of procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1 - Spectra Optia Followed by COBE Spectra | Arm 2 - COBE Spectra Followed by Spectra Optia
Number analyzed (Participants) | 17 | 15
minutes
  Spectra Optia Procedure Time | 136.8 (20.78) | 120.3 (17.58)
  COBE Spectra Procedure Time | 119.6 (18.65) | 112.3 (19.83)

9. Secondary Outcome: Usability/Assessment of System Operation - Adjustments
Description: Number of operator adjustments aimed at establishing and maintaining the plasma/ cellular interface: namely, on Spectra Optia, the adjustment of collection preference and, on COBE Spectra, the adjustment of the plasma pump flow rate.
Time Frame: Adjustments known immediately upon completion of the procedure
Measure: Mean (Standard Deviation); unit: number of adjustments
Arm/Group | Arm 1 - Spectra Optia Followed by COBE Spectra | Arm 2 - COBE Spectra Followed by Spectra Optia
Number analyzed (Participants) | 17 | 15
number of adjustments
  Spectra Optia adjustments | 4.6 (2.12) | 5.8 (2.48)
  COBE Spectra adjustments | 9.3 (3.67) | 10.7 (4.68)

10. Secondary Outcome: Usability/Assessment of System Operation - Device Malfunctions
Time Frame: Result know immediately upon successful completion of procedure
Measure: Number; unit: events
Groups:
- Spectra Optia vs COBE Spectra: All 32 subjects received both the Spectra Optia and the COBE Spectra. Device deficiency was not reported by randomization treatment arms.
Arm/Group | Spectra Optia vs COBE Spectra
Number analyzed (Participants) | 32
events
  Spectra Optia device deficiencies | 5
  COBE Spectra device deficiencies | 0

11. Secondary Outcome: Safety
Description: * Serious adverse events (SAEs) and unanticipated (serious) adverse device/procedure- related events (UADEs), adverse events (AEs).
  * any clinically significant changes to Complete Blood Count with differential white cell count (CBCD) and any significant changes to vital signs (temperature, heart rate, blood pressure) were captured as AEs. Also provided in full report to FDA.
Time Frame: 48-hours after last procedure
Measure: Number; unit: events
Arm/Group | Spectra Optia vs COBE Spectra
Number analyzed (Participants) | 32
events
  Spectra Optia SAEs | 0
  COBE Spectra SAEs | 0
  Spectra Optia UADEs | 0
  COBE Spectra UADEs | 0
  Number of subjects with >=1 AE | 17

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the point of randomization until 48-hours after the last study procedure.
Groups:
- Spectra Optia: A total of n=48 subjects were either randomized to receive a procedure (n=42) or were assigned the Spectra Optia as a lead-in subject (lead-in n=6). Lead-in donors were not randomized and received the Spectra Optia only for training purposes and are included for Spectra Optia safety only. Randomized subjects are included in safety regardless if they withdrew or did not complete a procedure. Spectra Optia events are AEs during the study period when the subject received the Spectra Optia.
- COBE Spectra: A total of n=42 subjects were randomized to receive a procedure. Randomized subjects are included in safety regardless if they withdrew or did not complete a procedure. Lead-in subjects are never exposed to COBE Spectra per protocol and not included. COBE Spectra events are AEs during the study period when the subject received the COBE Spectra.
Arm/Group | Spectra Optia | COBE Spectra
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/42
Other Adverse Events (participants affected / at risk) | 23/48 | 11/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spectra Optia (N=48) | COBE Spectra (N=42)
headache (Nervous system disorders) | 9 (10) | 6 (7) — expected due to mobilization medication
back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) — expected due to mobilization medication
insomnia (Psychiatric disorders) | 4 (4) | 2 (2) — expected due to mobilization medication
arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) — expected due to mobilization medication
haematoma (Vascular disorders) | 4 (4) | 0 (0) — expected related to venipuncture
sore shoulder (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
tingling (Nervous system disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The Full Analysis Set included 32 subjects who completed both procedures of the cross-over study design presented here. Two subjects did not meet pre-defined criteria for evaluable and 30 subjects were included in the Evaluable Analysis Population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less